CLINICAL TRIAL: NCT06809114
Title: A Phase I, First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of AT03-65 in Adults With Advanced Solid Tumors
Brief Title: FIH Study to Evaluate Safety, Tolerability, PK, PD & Preliminary Efficacy of AT03-65 With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Axcynsis Therapeutics Pte Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AT0365-P1-01
Record Dates: First submitted 2025-01-24; First posted 2025-02-05 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor

STUDY DESIGN:
Intervention Model Description: Dose escalation (Phase 1a) followed by Dose Expansion (Phase 1b)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AT03-65 Dose Escalation and Dose Expansion (Experimental): Subjects will receive AT03-65 via intravenous (IV) infusion on Day 1 of a 21-Day treatment cycle.
  Interventions: Drug: AT03-65

INTERVENTIONS:
Drug: AT03-65 — Treatment will continue until disease progression, unacceptable toxicity, subject withdrawal of consent or death.
  Other Names: AT03-65 Antibody Drug Conjugate

SUMMARY:
A Phase I, First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of AT03-65 in Adults with Advanced Solid Tumors

DETAILED DESCRIPTION:
This is a first-in-human (FIH), Phase 1, open-label, dose escalation and dose expansion study to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of AT03-65 in adults with advanced solid tumors. AT03-65 is administered via intravenous infusion using an accelerated escalation method for the lower 3 dose level groups and the 3 + 3 escalation method is used in the subsequent dose level groups.

The study design is to identify the maximum tolerated dose (MTD) and dose-limiting toxicities (DLT) during 21-day cycle. One or more doses or regimens lower than or at the MTD may be selected for further evaluations under Dose Expansion to further evaluate the IMP and identify the RP2D.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old at the time of signing written informed consent form (ICF).
2. Eastern cooperative oncology group (ECOG) Performance Status score of 0 or 1 at screening and on C1D1.
3. Pathologically documented, definitively diagnosed, advanced/metastatic solid tumor that is resistant or refractory to standard treatment, for which no further standard treatment is available, or the subject refuses or cannot tolerate standard therapy. Subjects must have measurable lesion according to response evaluation criteria in solid tumors (RECIST) v1.1.

3a) Monotherapy dose escalation study (Phase 1a):

* Subjects (with documented CLDN6 expression after the lower three dose levels) will be enrolled, including but not limited to the following histological subtypes: serous or endometrioid ovarian cancer, primary peritoneal cancer or fallopian tube cancer, endometrial cancer, NSCLC, breast cancer, esophageal cancer, and gastric/GEJ cancer. There is no upper limit on the number of prior treatment regimens the subject may have received.

  3b) Monotherapy cohort expansion study (Phase 1b)
* Subjects must meet the minimum requirement of CLDN6-expressing by IHC (cutoff value to be determined based on Phase Ia data and/or clinical studies of other CLDN6-targeting drugs), to be confirmed prior to enrollment.

Three cohorts will be involved:

Cohort 1: 24-30 subjects with advanced/metastatic CLDN6-expressing ovarian cancer, platinum resistant, refractory, or non-tolerant. Patients must have had one (or more) prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound, which may have included intraperitoneal therapy, high-dose therapy, consolidation, or extended therapy administered after completion of initial chemotherapy; patients must be considered platinum resistant or refractory according to standard Gynecologic Oncology Group (GOG) criteria, i.e., have had a treatment-free interval following platinum of 6 months or less, have persistent disease at the completion of primary platinum-based therapy or have progressed during platinum-based therapy, or be determined to be nontolerant after a recognized desensitization regimen.

Cohort 2: 24-30 subjects with advanced/metastatic CLDN6-expressing NSCLC. Subjects must have received at least one checkpoint inhibitor combination regimen (or platinum doublet where contraindicated). Patients with established driver mutations (epidermal growth factor receptor [EGFR], anaplastic lymphoma kinase [ALK], ROS proto-oncogene [ROS], mesenchymal epithelial transition factor [MET], rearranged during transfection [RET], B-Raf proto-oncogene, serine/threonine kinase [BRAF], and/or rat sarcoma [RAS]) must have progressed on standard of care for said mutation.

Cohort 3: 12 subjects with other advanced/metastatic CLDN6-expressing solid tumors who have exhausted options for standard of care therapies. There is no upper limit on the number of prior treatment regimens the subject may have received.

4) Subjects have fresh tumor sample or available archival block for CLDN6 IHC (except for the lower three dose levels of Phase Ia). If archival block samples from multiple timepoints are available, the most recent one is preferred.

5) Subjects with good organ function

6) Has a left ventricular ejection fraction (LVEF) ≥50% as determined by either an echocardiogram (ECHO) or multi-gated acquisition scan (MUGA) within 28 days before the start of study treatment.

7) Life expectancy ≥3 months.

8) Male subjects with female partners of childbearing potential and female subjects of childbearing potential must agree to use a highly effective form of contraception or avoid intercourse throughout the study period and for at least 6 months after the final administration of IMP. Males must agree not to freeze or donate sperm throughout the study period and for at least 6 months after final administration of IMP. Investigators will advise male subjects on the conservation of sperm prior to study treatment. Females must agree not to donate or retrieve ova for own use throughout the study period and for at least 6 months after final administration of IMP.

Exclusion Criteria:

1. Subjects previously received or is currently receiving any systemic anti-cancer therapy within 4 weeks or 5xT(1/2) if 5xT(1/2) of the drug/therapy used by the subject is confirmed to be < 4 weeks, 5xT(1/2) shall prevail] - prior to first dose of IMP
2. Not yet recovered to Grade 1 or baseline for treatment-related toxicities related to previous treatment with the exception of alopecia. The recovery time after surgery was less than 28 days
3. Subjects with clinically significant congenital or acquired cardiovascular diseases.
4. Presence of other active invasive cancers other than the one treated in this study within 5 years prior to screening, except appropriately treated BCC of the skin or in situ carcinoma of uterine cervix, or other local tumors considered cured by local treatment
5. Subjects with severe or uncontrolled systemic disease, including uncontrolled hypertension, uncontrolled diabetes mellitus, active bleeding diatheses, or active infection requiring intravenous injection (IV) of antibiotics, antivirals or antifungals
6. Subjects with medical history of clinically significant lung disease or who are suspected to have these disease by imagining at screening
7. Live vaccine within 4 weeks prior to first dose of IMP
8. Presence of active or untreated metastases to central nervous system or meninges or other evidence showing that metastatic lesions in central nervous system or meninges that have not yet been controlled at screening. Note: Subjects with central nervous system or meningeal metastases who are free of neurological symptoms not managed with steroids and stable by imagining 28 days after treatment prior to the first dose may be considered for enrollment
9. Presence of leptomeningeal disease.
10. Prior treatment with any ADC targeting CLDN6. Note: Prior treatment with immune engagers targeting CLDN6 is permitted.
11. Subjects who have received prior allogeneic or autologous bone marrow transplants.
12. Subjects who are pregnant (as confirmed by pregnancy tests performed within 7 days before enrollment) or planning to become pregnant.
13. Subjects who have received moderate or strong cytochrome P450 (CYP) 2C8 or CYP3A inhibitors or inducers, or P-glycoprotein (P-gp) inhibitors within 14 days prior to the first dose or cannot be discontinued during the study.
14. The investigator considers that the patient is not suitable for participating in this study (e.g.,IMP is not in the best interest of patient, patients with mental disorder, patients with poor compliance, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of AT03-65 | Up to 21 days
  The MTD is defined as the highest dose with an observed incidence of DLT in no more than one out of six patients treated at a particular dose level.
Dose-limiting toxicity (DLT) | Up to 21 days
  DLT refers to AEs that occurred during DLT observation period in dose escalation study, excluding toxicities clearly due to the underlying disease or extraneous causes.

SECONDARY OUTCOMES:
Determine levels of AT03-65 and its constituents over time in plasma | Maximum 2 years
  Assess PK concentration of AT03-65 in peripheral blood
Evaluate changes in circulating tumor DNA in plasma | Maximum 2 years
  Assess PD markers related to AT03-65 in peripheral blood
Determine the presence of antibodies to AT03-65 at different times in plasma | Maximum 2 years
  Assess immunogenicity concentration in peripheral blood
Assessment of Overall Response Rate (ORR) in subjects with advanced / metastatic solid tumors | Maximum 2 years
  Percentage of subjects whose best response is observed to be CR or PR throughout the study as assessed by local radiological assessment made by investigator according to RECIST V1.1
Determine the expression level of CLDN6 in tumor samples | Maximum 2 years
  Assess the presence and expression level of CLDN6 in tumor samples
Progress-Free Survival (PFS) of treatment in subjects with advanced / metastatic solid tumors | Maximum 2 years
  PFS as assessed by Local Investigators according to RECIST V1.1
Assessment of Disease Control Rate (DCR)in subjects with advanced / metastatic solid tumors | Maximum 2 years
  Percentage of subjects with best overall response of CR, PR and SD as assessed per RECIST v1.1
Assessment of Duration of Response (DOR) of treatment in patients with solid tumor | Maximum 2 years
  DOR as assessed by Local Investigators according to the RECIST V1.1
Assessment of Overall Survival (OS) of treatment in subjects with advanced / metastatic solid tumors | Maximum 2 years
  OS as assessed as duration from first dose of IMP to death
Assessment of Clinical Benefit Rate (CBR)in subjects with advanced / metastatic solid tumors | Maximum 2 years
  Percentage of subjects whose best response is observed to be CR, PR or SD

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University (OHSU), Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Data generated by this study will be considered confidential by the Investigator, except to the extent that it is included in a publication. The general strategy regarding publication of the study will be mutually agreed upon by the Investigator and Sponsor. The Sponsor reserves the right to manage the publication of all study results. The Investigator agrees that oral and written communication to third parties of any procedures or results from the study is subject to prior written consent of the Sponsor. Presentation material and/or manuscript(s) for publication will be reviewed by the Sponsor prior to submission for publication. Alterations in the material will only be made in agreement between the Investigator and the Sponsor